CLINICAL TRIAL: NCT02251275
Title: A Phase 3b, Multi-center, Open-label Trial to Evaluate the Long Term Safety of Immediate-release Tolvaptan (OPC-41061, 30 mg to 120 mg/Day, Split Dose) in Subjects With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Long Term Safety of Immediate-release Tolvaptan in Subjects With Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-13-211
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tolvaptan (Experimental): Tolvaptan was self-administered orally as split-dose regimens. The dose regimens used in this trial were 15/15 milligram (mg), 30/15 mg, 45/15 mg, 60/30 mg, or 90/30 mg. Starting doses were dependent upon the participant's previous trial as follows:
  * Trial 156-13-210: initiated on tolvaptan at a split-dose of 45/15 mg with upward titration every 3 to 4 days to 60/30 mg or 90/30 mg per day according to tolerability.
  * Trial 156-08-271: retained the last dose level of tolvaptan received in the trial (45/15 mg, 60/30 mg, or 90/30 mg) and started at that same dose in Trial 156-13-211.
  * Other Trials (156-04-251 and 156-09-290): initiated on tolvaptan at a split-dose of 45/15 mg with upward titration every 3 to 4 days to 60/30 mg or 90/30 mg per day according to tolerability.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan tablets (15 or 30 mg) self-administered orally as split-dose regimens, once upon awakening and another approximately 8 to 9 hours later
  Other Names: OPC-41061

SUMMARY:
The purpose of the trial was to evaluate and describe the long term safety of tolvaptan in participants with autosomal dominant polycystic kidney disease (ADPKD).

DETAILED DESCRIPTION:
This was a Phase 3b trial to evaluate and describe the long term safety of tolvaptan treatment in ADPKD participants with chronic kidney disease (CKD). Eligible participants could enroll into Trial 156-13-211 after completing the follow-up visit(s) of their previous trial (156-13-210, 156-08-271, 156-04-251, or 156-09-290). Renal function was assessed during screening by using historical laboratory values for serum creatinine levels to calculate the estimated glomerular filtration rate (eGFR).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 years with confirmed diagnosis of ADPKD (during participation in prior tolvaptan trials) who have completed and transferred from the double-blind Trial 156-13-210 (12-month period including post treatment follow-up, regardless of whether this was on-treatment or off-treatment), or completed Trial 156-08-271 or a prior tolvaptan trial, or interrupted or discontinued treatment in a prior tolvaptan ADPKD trial other than Trial 156-13-210. Participants may be enrolled with the medical monitor approval, and additional close monitoring may be required at the beginning of the trial.
* eGFR ≥ 20 milliliter (mL)/minute (min)/1.73 meter squared (m^2) within 3 months prior to the baseline visit. Participants who have an eGFR ≤ 20 mL/min/1.73 m^2 may be enrolled with medical monitor approval.

Exclusion Criteria:

* Need for chronic diuretic use
* Hepatic impairment based on liver function abnormalities other than that expected for ADPKD with cystic liver disease
* Women of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of investigational medicinal product (IMP)
* Women who are breast-feeding and/or who have a positive pregnancy test result prior to receiving IMP.
* Participants with contraindications to required trial assessments (contraindications to optional assessments, for example, magnetic resonance imaging [MRI] are not a limitation).
* Participants who in the opinion of the investigator or the medical monitor, have a medical history or medical finding inconsistent with safety or trial compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1803 (Actual)
Dates: Start 2014-10-17 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (185):
- United States (73):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Stanford, California
  - Aurora, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Hudson, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Ocala, Florida
  - Port Charlotte, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Meridian, Idaho
  - Chicago, Illinois
  - Kansas City, Kansas
  - Wichita, Kansas
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Greenbelt, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Pontiac, Michigan
  - Roseville, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Reno, Nevada
  - Eatontown, New Jersey
  - Voorhees Township, New Jersey
  - Buffalo, New York
  - Laurelton, New York
  - Mineola, New York
  - New York, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Doylestown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - McAllen, Texas
  - Burlington, Vermont
  - Arlington, Virginia
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Wenatchee, Washington
  - Morgantown, West Virginia
- Argentina (5):
  - Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Junín, Buenos Aires
  - Pergamino, Buenos Aires
  - Pilar, Buenos Aires
  - Córdoba
- Australia (11):
  - Camperdown, New South Wales
  - New Lambton Heights, New South Wales
  - St Leonards, New South Wales
  - Westmead, New South Wales
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Launceston, Tasmania
  - Parkville, Victoria
  - Reservoir, Victoria
  - Richmond, Victoria
  - Perth, Western Australia
- Belgium (7):
  - Aalst
  - Brussels
  - Edegem
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
- Canada (5):
  - Edmonton, Alberta
  - Mount Pearl, Newfoundland and Labrador
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (8):
  - Brno
  - České Budějovice
  - Hradec Králové
  - Jihlava
  - Jilemnice
  - Liberec
  - Ostrava
  - Prague
- Denmark (3):
  - Aalborg
  - Aarhus N
  - Holstebro
- Germany (8):
  - Heidelberg, Baden-Wurttemberg
  - Munich, Bavaria
  - Nuremberg, Bavaria
  - Wiesbaden, Hesse
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Dresden, Saxony
  - Berlin
- Hungary (3):
  - Budapest
  - Pécs
  - Szeged
- Israel (6):
  - Ashkelon
  - Jerusalem
  - Nahariya
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (7):
  - Montichiari, Brescia
  - Bari
  - Lecco
  - Milan
  - Modena
  - Napoli
  - Pavia
- Netherlands (3):
  - Amsterdam
  - Groningen
  - Nijmegen
- Bergen, Norway
- Poland (9):
  - Ciechanów
  - Gdansk
  - Golub-Dobrzyń
  - Krakow
  - Lodz
  - Lublin
  - Szczecin
  - Warsaw
  - Wroclaw
- Romania (2):
  - Bucharest
  - Oradea
- Russia (4):
  - Kemerovo
  - Krasnoyarsk
  - Saint Petersburg
  - Yaroslavl
- South Africa (3):
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
- Spain (4):
  - Barcelona
  - Ciudad Real
  - Madrid
  - Valencia
- Sweden (4):
  - Gothenburg
  - Linköping
  - Stockholm
  - Uppsala
- United Kingdom (19):
  - Belfast, County Antrim
  - Exeter, Devon
  - Hull, East Riding Of Yorkshire
  - Brighton, East Sussex
  - London, Greater London
  - Manchester, Greater Manchester
  - Salford, Greater Manchester
  - Stevenage, Hertfordshire
  - Inverness, Highland Region
  - Leicester, Leicestershire
  - Edinburgh, Lothian Region
  - Liverpool, Norfolk
  - Sheffield, South Yorkshire
  - Stoke-on-Trent, Staffordshire
  - Newcastle upon Tyne, Tyne & Wear
  - Coventry, Warwickshire
  - Birmingham, West Midlands
  - Middlesbrough
  - Swansea

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com

REFERENCES:
- [Derived] Chebib FT, Zhou X, Garbinsky D, Davenport E, Nunna S, Oberdhan D, Fernandes A. Tolvaptan and Kidney Function Decline in Older Individuals With Autosomal Dominant Polycystic Kidney Disease: A Pooled Analysis of Randomized Clinical Trials and Observational Studies. Kidney Med. 2023 Apr 14;5(6):100639. doi: 10.1016/j.xkme.2023.100639. eCollection 2023 Jun. PMID 37250503
- [Derived] Alpers DH, Lewis JH, Hunt CM, Freston JW, Torres VE, Li H, Wang W, Hoke ME, Roth SE, Westcott-Baker L, Estilo A. Clinical Pattern of Tolvaptan-Associated Liver Injury in Trial Participants With Autosomal Dominant Polycystic Kidney Disease (ADPKD): An Analysis of Pivotal Clinical Trials. Am J Kidney Dis. 2023 Mar;81(3):281-293.e1. doi: 10.1053/j.ajkd.2022.08.012. Epub 2022 Sep 30. PMID 36191725
- [Derived] Torres VE, Chapman AB, Devuyst O, Gansevoort RT, Perrone RD, Lee J, Hoke ME, Estilo A, Sergeyeva O. Multicenter Study of Long-Term Safety of Tolvaptan in Later-Stage Autosomal Dominant Polycystic Kidney Disease. Clin J Am Soc Nephrol. 2020 Dec 31;16(1):48-58. doi: 10.2215/CJN.10250620. Epub 2020 Dec 29. PMID 33376102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants could enroll into Trial 156-13-211 after completing follow-up visit(s) of their previous trial (156-13-210, 156-08-271, 156-04-251, or 156-09-290).
Pre-assignment Details: One participant screened, but withdrew consent on the same day (prior to study drug treatment) and is not included in the study data.
  Starting doses depended on the participant's previous trial.
Groups:
- Tolvaptan (From 156-13-210: Tolvaptan): Participants were previously treated with tolvaptan in Trial 156-13-210. Participants initiated on tolvaptan at a split-dose of 45/15 milligrams (mg) with upward titration every 3 to 4 days to 60/30 mg or 90/30 mg per day according to tolerability.
- Tolvaptan (From 156-13-210: Placebo): Participants were previously treated with placebo in Trial 156-13-210. Participants initiated on tolvaptan at a split-dose of 45/15 mg with upward titration every 3 to 4 days to 60/30 mg or 90/30 mg per day according to tolerability.
- Tolvaptan (From 156-08-271: Tolvaptan): Participants were previously treated with tolvaptan in Trial 156-08-271. Participants retained the last dose level of tolvaptan received in the trial (45/15 mg, 60/30 mg, or 90/30 mg) and started at that same dose in Trial 156-13-211.
- Tolvaptan (From Other: Tolvaptan): Participants were previously treated with tolvaptan in Other Trials (156-04-251 and 156-09-290). Participants initiated on tolvaptan at a split-dose of 45/15 mg with upward titration every 3 to 4 days to 60/30 mg or 90/30 mg per day according to tolerability.
- Tolvaptan (From Other: Placebo): Participants were previously treated with placebo in Other Trials (156-04-251 and 156-09-290). Participants initiated on tolvaptan at a split-dose of 45/15 mg with upward titration every 3 to 4 days to 60/30 mg or 90/30 mg per day according to tolerability.
Period: Overall Study
Arm/Group | Tolvaptan (From 156-13-210: Tolvaptan) | Tolvaptan (From 156-13-210: Placebo) | Tolvaptan (From 156-08-271: Tolvaptan) | Tolvaptan (From Other: Tolvaptan) | Tolvaptan (From Other: Placebo)
Started | 506 | 570 | 718 | 6 (From trials 156-04-251 and 156-09-290) | 3 (From trials 156-04-251 and 156-09-290)
Received at Least 1 Dose of Study Drug | 505 | 569 | 717 | 6 | 3
Completed | 434 | 423 | 624 | 5 | 2
Not Completed | 72 | 147 | 94 | 1 | 1
Not completed — Adverse Event | 23 | 60 | 28 | 0 | 0
Not completed — Lost to Follow-up | 5 | 6 | 4 | 0 | 0
Not completed — Physician Decision | 19 | 30 | 26 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 51 | 35 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who enrolled in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan (From 156-13-210: Tolvaptan) | Tolvaptan (From 156-13-210: Placebo) | Tolvaptan (From 156-08-271: Tolvaptan) | Tolvaptan (From Other: Tolvaptan) | Tolvaptan (From Other: Placebo) | Total
Number analyzed (Participants) | 506 | 570 | 718 | 6 | 3 | 1803
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.9 (8.1) | 48.6 (8.0) | 45.5 (7.8) | 41.2 (11.4) | 47.0 (2.6) | 47.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 290 | 343 | 5 | 2 | 874
  Male | 272 | 280 | 375 | 1 | 1 | 929
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 25 | 49 | 1 | 0 | 102
  Not Hispanic or Latino | 479 | 545 | 669 | 5 | 3 | 1701
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 0 | 0 | 3
  Asian | 16 | 16 | 10 | 0 | 0 | 42
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 0 | 0 | 3
  Black or African American | 19 | 23 | 6 | 0 | 0 | 48
  White | 461 | 525 | 694 | 6 | 3 | 1689
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 6 | 0 | 0 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was as any untoward medical occurrence associated with the use of an investigational medicinal product (IMP), whether or not considered IMP related. A TEAE was an AE that started after trial drug treatment; or if the event was continuous from baseline and was serious, related to IMP, or resulted in death, discontinuation, interruption or reduction of trial therapy. A serious TEAE included any event that resulted in: death, life-threatening, persistent or significant incapacity, substantial disruption of ability to conduct normal life functions, required inpatient hospitalization, prolonged hospitalization, congenital anomaly/birth defect, or other medically significant events as per medical judgment, that jeopardized the participant and that required medical or surgical intervention. A severe TEAE was an inability to work or perform normal daily activity. A summary of serious and all other non-serious TEAEs, regardless of causality, is located in the AE section.
Time Frame: Baseline through end of treatment (up to 42 months) and follow-up 7 days posttreatment(+ 7 days)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tolvaptan (From 156-13-210: Tolvaptan) | Tolvaptan (From 156-13-210: Placebo) | Tolvaptan (From 156-08-271: Tolvaptan) | Tolvaptan (From Other: Tolvaptan) | Tolvaptan (From Other: Placebo)
Number analyzed (Participants) | 505 | 569 | 717 | 6 | 3
participants
  Participants with TEAEs | 473 | 531 | 640 | 6 | 3
  Participants with serious TEAEs | 87 | 96 | 103 | 1 | 2
  Participants with severe TEAEs | 74 | 78 | 83 | 2 | 1
  Discontinued due to TEAEs | 33 | 65 | 38 | 0 | 1
  Deaths | 1 | 5 | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through end of treatment (up to 42 months) and follow-up 7 days posttreatment (+ 7 days)
Arm/Group | Tolvaptan (From 156-13-210: Tolvaptan) | Tolvaptan (From 156-13-210: Placebo) | Tolvaptan (From 156-08-271: Tolvaptan) | Tolvaptan (From Other: Tolvaptan) | Tolvaptan (From Other: Placebo)
All-Cause Mortality (participants affected / at risk) | 1/505 | 5/569 | 3/717 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 87/505 | 96/569 | 103/717 | 1/6 | 2/3
Other Adverse Events (participants affected / at risk) | 469/505 | 525/569 | 633/717 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tolvaptan (From 156-13-210: Tolvaptan) (N=505) | Tolvaptan (From 156-13-210: Placebo) (N=569) | Tolvaptan (From 156-08-271: Tolvaptan) (N=717) | Tolvaptan (From Other: Tolvaptan) (N=6) | Tolvaptan (From Other: Placebo) (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral Valve Prolapse (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Ventricular Dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Aortic Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polycystic Liver Disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urachal Abnormality (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Borderline Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocrine Ophthalmopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Cyst Infection (Infections and infestations) | 5 (7) | 8 (10) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cat Scratch Disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cyst Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster Oticus (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infected Cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirenal Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous Fistula Site Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anastomotic Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour Marker Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver Function Test Increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
International Normalised Ratio Fluctuation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Glomerular Filtration Rate Decreased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Urine Present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma of Head and Neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/272 (1) | 1/280 (1) | 0/375 (0) | 0/1 (0) | 0/1 (0) — The adverse event occurs in only male participants.
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian Theca Cell Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/234 (0) | 1/290 (1) | 0/343 (0) | 0/5 (0) | 0/1 (0) — The adverse event occurs in only female participants.
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carcinoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to Adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-Cell Small Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ruptured Cerebral Aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vith Nerve Paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basilar Artery Aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar Ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Pain (Renal and urinary disorders) | 2 (2) | 5 (7) | 1 (1) | 0 (0) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 6 (6) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Renal Haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Renal Cyst Haemorrhage (Renal and urinary disorders) | 3 (4) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Cyst Ruptured (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 5 (5) | 8 (9) | 7 (7) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Kidney Enlargement (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
End Stage Renal Disease (Renal and urinary disorders) | 3 (3) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1/234 (1) | 0/290 (0) | 0/343 (0) | 0/5 (0) | 0/2 (0) — The adverse event occurs in only female participants.
Breast Enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0/234 (0) | 1/290 (1) | 0/343 (0) | 0/5 (0) | 0/2 (0) — The adverse event occurs in only female participants.
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Laxity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteritis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aortic Dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tolvaptan (From 156-13-210: Tolvaptan) (N=505) | Tolvaptan (From 156-13-210: Placebo) (N=569) | Tolvaptan (From 156-08-271: Tolvaptan) (N=717) | Tolvaptan (From Other: Tolvaptan) (N=6) | Tolvaptan (From Other: Placebo) (N=3)
Left Ventricular Hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 5 (5) | 6 (6) | 14 (15) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Motion Sickness (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 9 (10) | 14 (16) | 4 (5) | 1 (1) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 7 (7) | 1 (1) | 6 (6) | 0 (0) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 6 (6) | 6 (7) | 6 (6) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 20 (24) | 19 (24) | 12 (12) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (17) | 28 (34) | 10 (11) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 37 (41) | 38 (43) | 33 (39) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 22 (24) | 38 (41) | 3 (4) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 17 (19) | 27 (28) | 10 (10) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 11 (11) | 19 (22) | 17 (17) | 0 (0) | 1 (1)
Gingival Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 37 (40) | 51 (59) | 38 (40) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 24 (27) | 38 (41) | 32 (36) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 47 (55) | 74 (85) | 34 (37) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 5 (5) | 5 (5) | 4 (4) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 32 (37) | 39 (46) | 42 (49) | 0 (0) | 0 (0)
Pain (General disorders) | 6 (9) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Thirst (General disorders) | 139 (176) | 183 (213) | 91 (99) | 4 (4) | 0 (0)
Type I Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 23 (25) | 29 (34) | 31 (35) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 8 (9) | 9 (9) | 5 (8) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 14 (15) | 22 (24) | 41 (44) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 34 (38) | 43 (49) | 39 (52) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 92 (129) | 100 (143) | 94 (123) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 22 (30) | 31 (37) | 35 (47) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 58 (64) | 53 (83) | 86 (129) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 52 (86) | 58 (79) | 65 (117) | 1 (1) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 3/234 (3) | 1/290 (1) | 6/343 (7) | 0/5 (0) | 1/2 (1) — The adverse event occurs in only female participants.
Zika Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (10) | 9 (10) | 11 (11) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 7 (9) | 19 (26) | 17 (21) | 1 (1) | 0 (0)
Blood Calcium Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 77 (104) | 87 (129) | 69 (87) | 0 (0) | 1 (1)
Kidney Palpable (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 4 (4) | 5 (6) | 2 (3) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 3 (3) | 4 (5) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 8 (9) | 18 (19) | 4 (4) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 28 (49) | 25 (46) | 30 (42) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (5) | 5 (5) | 7 (7) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 27 (29) | 53 (54) | 14 (14) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (42) | 25 (26) | 26 (36) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 53 (59) | 57 (71) | 51 (55) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 18 (20) | 31 (37) | 31 (37) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 51 (61) | 72 (83) | 51 (68) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 9 (9) | 9 (9) | 13 (15) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 4 (4) | 6 (6) | 7 (7) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 27 (34) | 52 (63) | 48 (53) | 0 (0) | 2 (2)
Nocturia (Renal and urinary disorders) | 77 (105) | 124 (150) | 58 (63) | 3 (4) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 27 (36) | 34 (38) | 12 (18) | 2 (2) | 0 (0)
Polyuria (Renal and urinary disorders) | 117 (141) | 180 (203) | 53 (56) | 2 (2) | 0 (0)
Renal Cyst Ruptured (Renal and urinary disorders) | 4 (4) | 9 (12) | 7 (8) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 12 (12) | 29 (31) | 14 (16) | 0 (0) | 0 (0)
Renal Pain (Renal and urinary disorders) | 98 (139) | 110 (179) | 141 (209) | 3 (4) | 2 (3)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0/234 (0) | 1/290 (1) | 3/343 (3) | 0/5 (0) | 1/2 (1) — The adverse event occurs in only female participants.
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (30) | 27 (31) | 28 (31) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 7 (9) | 4 (5) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 87 (116) | 77 (97) | 139 (163) | 4 (4) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2015-03-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT02251275/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT02251275/SAP_001.pdf